CLINICAL TRIAL: NCT05274425
Title: A 24-week Prospective, Open-label, Multicenter, Single-arm, Observational Regulatory Post-Marketing Surveillance (rPMS) Study in Real-world Setting (Mandatory by Local HA Regulation) for Enerzair (QVM149 150/50/80 μg o.d. and QVM149 150/50/160 μg o.d. Via Breezhaler)
Brief Title: A 24-week rPMS Study in Real-world Setting for Enerzair
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CQVM149BKR01
Record Dates: First submitted 2021-11-30; First posted 2022-03-10 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Asthma
Keywords: Enerzair; QVM149; Korea
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Enerzair 150/50/80 μg: Enerzair inhalation capsule (indacaterol acetate/glycopyrronium bromide/mometasone furoate; 150/50/80 μg) via Breezhaler
  Interventions: Other: Enerzair 150/50/80 μg
- Enerzair 150/50/160 μg: Enerzair inhalation capsule (indacaterol acetate/glycopyrronium bromide/mometasone furoate; 150/50/160 μg) via Breezhaler,
  Interventions: Other: Enerzair 150/50/160 μg

INTERVENTIONS:
Other: Enerzair 150/50/80 μg — There is no treatment allocation. Patients administered Enerzair by prescription that have started before inclusion of the patient into the study will be enrolled.
  Groups: Enerzair 150/50/80 μg
Other: Enerzair 150/50/160 μg — There is no treatment allocation. Patients administered Enerzair by prescription that have started before inclusion of the patient into the study will be enrolled.
  Groups: Enerzair 150/50/160 μg

SUMMARY:
This surveillance was designed as a prospective, open-label, multicenter, single-arm, non-interventional, observational study to evaluate the safety and effectiveness of Enerzair inhalation capsule for up to 24 weeks under routine clinical practice.

DETAILED DESCRIPTION:
The two different doses of Enerzair inhalation capsule via Breezhaler will be prescribed according to the approved label information in Korea, and the investigation for any additional diagnostic or monitoring will be not conducted for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years of age) with a physician's diagnosis of asthma, who are prescribed Enerzair inhalation capsule (indacaterol acetate/ glycopyrronium bromide/mometasone furoate; 150/50/80, 150/50/160 μg) via Breezhaler, as per the approved label information
2. Patients who participate in the study after signing the consent form for data collection and use (Data Privacy ICF) after receiving a clear explanation of the objectives and nature of the study from the investigator

Exclusion Criteria:

1. Patients who are contraindicated for this medicinal product as described in the Precautions for Use in the label information (package insert) A. Patients with hypersensitivity reaction to this medicinal product or any of its constituents B. Because this medicinal product contains lactose, patients with hereditary problems of galactose intolerance, the Lapp lactose deficiency or glucose-galactose malabsorption, etc.
2. Patients with acute asthma symptoms, including acute episodes of bronchospasm, for which a short-acting bronchodilator is required
3. Patients participating in other interventional clinical trials

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who received at least one dose of Enerzair inhalation capsule via Breezhaler and that have provided consent for their data collection.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2027-03-11 (Estimated); Study Completion 2027-03-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | 24 weeks
  Incidence of AE and SAE to be collected
Incidence of unexpected adverse events and unexpected serious adverse events | 24 weeks
  Incidence of unexpected AE and SAE. The term "unexpected" means not listed in local label.

SECONDARY OUTCOMES:
Change from baseline in trough FEV1 | Baseline, week 12
  Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer.
Change from baseline in ACT score | Baseline, week 12
  The Asthma Control Test (ACT) is a validated tool to assess overall asthma control. It is a 1 page questionnaire consisting of 5 simple questions assessing: asthma symptoms, use of rescue medications, and the impact of asthma on everyday functioning. All questions are scored on a 5-point Likert scale, with a higher score indicating better control. All scores are added together to calculate a total score. Total score ranges from 5 to 25. A positive change indicates improvement.
Effective rate and ineffective rate by investigator assessment | week 12
  The investigator comprehensively and subjectively evaluates the therapeutic effect of a treatment.
  The investigators can select effective, if they think patient's symptom was improved or ineffective, if they think patient's symptom was unchanged/aggravated.
Baseline characteristics of patients showing adverse events | 24 weeks
  The incidence rates of AEs will be presented by factors, such as subject baseline characteristics (age (<65 vs. ≥65 years), male vs. female, pregnancy (yes vs. no), family history (yes vs. no), exacerbation history (0 vs. above 1), smoking history (yes vs. no), comorbidity (yes vs. no), concomitant medication/ therapy (yes vs. no)), study treatment information, and special populations.
Baseline characteristics of patients showing adverse drug reactions | 24 weeks
  The incidence rates of ADRs will be presented by factors, such as subject baseline characteristics (age (<65 vs. ≥65 years), male vs. female, pregnancy (yes vs. no), family history (yes vs. no), exacerbation history (0 vs. above 1), smoking history (yes vs. no), comorbidity (yes vs. no), concomitant medication/ therapy (yes vs. no)), study treatment information, and special populations.
Baseline characteristics of patients in relation to changes from baseline in trough FEV1 | 12 weeks
  Regression analysis will be performed to determine factors affecting the change in trough FEV1, out of baseline characteristics (age (<65 vs. ≥65 years), male vs. female, pregnancy (yes vs. no), family history (yes vs. no), exacerbation history (0 vs. 1), smoking history (yes vs. no), comorbidity (yes vs. no), concomitant medication/ therapy (yes vs. no)), study treatment information, and special populations.
Baseline characteristics of patients in relation to changes from baseline in trough ACT score | 12 weeks
  Regression analysis will be performed to determine factors affecting the change in trough ACT score, out of baseline characteristics (age (<65 vs. ≥65 years), male vs. female, pregnancy (yes vs. no), family history (yes vs. no), exacerbation history (0 vs. 1), smoking history (yes vs. no), comorbidity (yes vs. no), concomitant medication/ therapy (yes vs. no)), study treatment information, and special populations.
Baseline characteristics of patients in relation to the investigator assessment | 12 weeks
  Logistic regression analysis will be performed to determine factors affecting the effectiveness (improved) in the investigator assessment, out of baseline characteristics (age (<65 vs. ≥65 years), male vs. female, pregnancy (yes vs. no), family history (yes vs. no), exacerbation history (0 vs. above 1), smoking history (yes vs. no), comorbidity (yes vs. no), concomitant medication/ therapy (yes vs. no)), study treatment information, and special populations.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- South Korea (13):
  - Novartis Investigative Site, Daegu, Dalseo Gu
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Deogyang Gu Goyang Si, Gyeonggi-do
  - Novartis Investigative Site, Jeonju, Jeollabuk-do
  - Novartis Investigative Site, Suncheon, Jeollanam-do
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Gyeongsangnam Do
  - Novartis Investigative Site, Seoul

IPD SHARING:
Plan to Share IPD: No